CLINICAL TRIAL: NCT04691310
Title: The Efficacy of Kinesio Taping on Neck Lymphedema Following Head and Neck Cancer Therapy: Double Blind Randomized Placebo Controlled Study
Brief Title: The Efficacy of Kinesio Taping on Lymphedema Following Head and Neck Cancer Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Sevgi Atar, Medical Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 309, 2020-082
Record Dates: First submitted 2020-12-26; First posted 2020-12-31 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Lymphedema; Head and Neck Cancer; Kinesio Taping; Therapy
Keywords: Kinesio taping; neck; lymphedema; head; cancer; therapy
MeSH Terms: conditions — Lymphedema; Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Kinesio taping study (Active Comparator): Kinesio tex gold tape was applied to neck localised lymphedema as stretched. Kinesio tape maintained during consecutive days and also were re applied with manual lymphatic drainage therapy as 5 times first week, and afterthat 2 times for 3 weeks (total 4 weeks)
  Interventions: Device: Kinesio Tex Gold
- Kinesio taping sham (Sham Comparator): Kinesio tex gold tape was applied to neck localised lymphedema as no-stretched. Kinesio tape maintained during consecutive days and also were re applied with manual lymphatic drainage therapy as 5 times first week, and afterthat 2 times for 3 weeks (total 4 weeks)
  Interventions: Device: Kinesio Tex Gold

INTERVENTIONS:
Device: Kinesio Tex Gold — The Kinesio Tex Gold is a kinesio tape that had been certified and patented.

SUMMARY:
Purpose off the study is investigating to efficacy of kinesio taping on neck lymphedema after the head and neck cancer therapy.

DETAILED DESCRIPTION:
The neck lymphedema is a multidirectional process that depends on lymphatic circulation issues. The lymphedema can be treated using such as therapies, drugs or surgeries. There are few techniques for treatment of neck lymphedema and also in our best knowledge the kinesio taping therapy on lymphedema following neck cancer therapy had not been investigated or published. The study will assess the efficacy of kinesio taping in neck lymphedema with manual therapy after the head and neck cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years
* External neck lymphedema
* Head and neck cancer treatment patients
* patients who have not open wound on neck
* Patients who were accept to consent form

Exclusion Criteria:

* Mental disorders Cognitive limitations Pregnancy Out of age 18-70 years old Patients who were not accept to consent form

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The values of diameter of lymphedema of neck with face | Baseline
  The diameters of upper, middle and lower points of neck were measured with tailor meter by a Physical Medicine and Rehabilitation professionals (measure unit is cm).
The values of diameter of lymphedema of neck with face | 2 weeks
  The diameters of upper, middle and lower points of neck and two points of face were measured with tailor meter by a Physical Medicine and Rehabilitation professionals (measure unit is cm).
The values of diameter of lymphedema of neck with face | 4 weeks
  The diameters of upper, middle and lower points of neck and two points of face were measured with tailor meter by a Physical Medicine and Rehabilitation professionals (measure unit is cm). The changes were assessed from baseline neck diameter at end of treatment and after one month.
The values of diameter of lymphedema of neck with face | 8 weeks
  The diameters of upper, middle and lower points of neck were measured with tailor meter by a Physical Medicine and Rehabilitation professionals (measure unit is cm). The changes were assessed from baseline neck diameter at end of treatment and after one month.
The outcomes of Quality of Life Questionnaire-Head and Neck 35 | baseline
  It was assessed by Quality of Life Questionnaire-Head and Neck 35 that a self questionnaire in head and neck cancer patients. The minimum score is 0 and maximum score is 100. The high scores were worst low scores were good health.
The outcomes of Quality of Life Questionnaire-Head and Neck 35 | 4 weeks
  It was assessed by Quality of Life Questionnaire-Head and Neck 35 that a self questionnaire in head and neck cancer patients. The minimum score is 0 and maximum score is 100. The high scores were worst low scores were good health.
The outcomes of Quality of Life Questionnaire-Head and Neck 35 | 8 weeks
  It was assessed by Quality of Life Questionnaire-Head and Neck 35 that a self questionnaire in head and neck cancer patients. The minimum score is 0 and maximum score is 100. The high scores were worst low scores were good health.
The scores of head and neck external lymphedema rating scale | Baseline
  They were assessed by M. D. Anderson head and neck lymphedema rating scale in head and neck cancer patients. Composite Score ranges from 0 ( low edema) to 3 (high level edema).
The scores of head and neck external lymphedema rating scale | 2 weeks
  They were assessed by M. D. Anderson head and neck lymphedema rating scale in head and neck cancer patients. Composite Score ranges from 0 ( low edema) to 3 (high level edema).
The scores of head and neck external lymphedema rating scale | 4 weeks
  They were assessed by M. D. Anderson head and neck lymphedema rating scale in head and neck cancer patients. Composite Score ranges from 0 ( low edema) to 3 (high level edema).
The scores of head and neck external lymphedema rating scale | 8 weeks
  They were assessed by M. D. Anderson head and neck lymphedema rating scale in head and neck cancer patients. Composite Score ranges from 0 ( low edema) to 3 (high level edema).
The outcomes of Patterson larynx pharynx internal edema scale | Baseline
  It was assessed with Flexible Endoscopic Evaluation Study. Flexible Endoscopic Evaluation Study results were scored on Patterson larynx pharynx edema scale. The scores of scale were no, mild, moderate and severe . The high grade symptom scores were worst, low scores were good health
The outcomes of Patterson larynx pharynx edema scale | 2 weeks
  It was assessed with Fiberoptic Endoscopic Evaluation Study. Flexible Endoscopic Evaluation Study results were scored on Patterson larynx pharynx edema scale. The scores of scale were no, mild, moderate and severe. The high grade symptom scores were worst, low scores were good health
The outcomes of Patterson larynx pharynx edema scale | 4 weeks
  It was assessed with Fiberoptic Endoscopic Evaluation Study. Flexible Endoscopic Evaluation Study results were scored on Patterson larynx pharynx edema scale. The scores of scale were no, mild, moderate and severe. The high grade symptom scores were worst, low scores were good health
The outcomes of Patterson larynx pharynx edema scale | 8 weeks
  It was assessed with Fiberoptic Endoscopic Evaluation Study. Flexible Endoscopic Evaluation Study results were scored on Patterson larynx pharynx edema scale. The scores of scale were no, mild, moderate and severe. The high grade symptom scores were worst, low scores were good health

SECONDARY OUTCOMES:
Mean of demographic | Baseline
  Age, gender, history of smoke, history of morbidities, diagnosis, stage, therapies of cancer, lymphedema stages were noted

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Atar, Special.,MD, Study Director — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasawara KT, Mapa JMR, Ferreira V, Added MAN, Shiwa SR, Carvas N Jr, Batista PA. Effects of Kinesio Taping on breast cancer-related lymphedema: A meta-analysis in clinical trials. Physiother Theory Pract. 2018 May;34(5):337-345. doi: 10.1080/09593985.2017.1419522. Epub 2018 Jan 8. PMID 29308967
- [Background] Deng J, Murphy BA, Dietrich MS, Wells N, Wallston KA, Sinard RJ, Cmelak AJ, Gilbert J, Ridner SH. Impact of secondary lymphedema after head and neck cancer treatment on symptoms, functional status, and quality of life. Head Neck. 2013 Jul;35(7):1026-35. doi: 10.1002/hed.23084. Epub 2012 Jul 12. PMID 22791550